CLINICAL TRIAL: NCT05147285
Title: The Effect of Different Exercise Modalities Applied by Tele Rehabilitation on Functional Capacity, Oxidative Stress and Respiratory Parameters in Cystic Fibrosis Children
Brief Title: The Effect of Telerehabilitation on Functional Capacity, Oxidative Stress and Respiratory Parameters in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kübra Kılıç, Physiotherapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-20069
Record Dates: First submitted 2021-10-31; First posted 2021-12-07 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Cystic Fibrosis; Telerehabilitation
Keywords: exercise; oxidative stress; respiratory muscles
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stabilization group (Experimental): Only stabilization exercises in patients with cystic fibrosis
  Interventions: Other: stabilization exercises
- combined group (Experimental): stabilization exercise and aerobic exercise training in patients with cystic fibrosis
  Interventions: Other: combined exercises
- control group (Experimental): physical activity recommendations in patients with cystic fibrosis
  Interventions: Other: Physical activity recommendations

INTERVENTIONS:
Other: stabilization exercises — Patients will be applied only online supervised stabilization exercises three times a week for 8 weeks.
  Arms: Stabilization group
Other: combined exercises — Patients will be applied online supervised aerobic exercise training and stabilization exercises.Aerobic exercises will be performed for 8 weeks, for 30-45 minutes, at 65-75% of the maximum heart rate, 3 days a week, on the days when stabilization exercises are not performed.
  Arms: combined group
Other: Physical activity recommendations — The importance of physical activity will be explained to the patients and appropriate physical activity recommendations will be made.
  Arms: control group

SUMMARY:
The aim of this study is to examine the effects of different exercise modalities applied with tele-rehabilitation on functional capacity, oxidative stress and respiratory parameters in children with cystic fibrosis

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most common life-shortening autosomal recessive disease among populations of caucasians with a frequency of 1 in 2000 to 3000 live births. The most common problems in these patients are increased bronchial secretion, decreased exercise capacity, and shortness of breath. In addition to progressive respiratory disease, peripheral and respiratory muscle function impairments, inflammation, and contribute to the decrease in exercise capacity in CF patients. Recent studies show that increased oxidative stress and impaired oxidant / antioxidant capacity have an important role in disease progression in CF patients. CF childrens may be more physically inactive. Cystic fibrosis transmembrane regulator (CFTR) modulators, airway clearance therapies, chest physiotherapy and exercise trainings are treatment options in these populations. Regular exercise which is the component of pulmonary rehabilitation (PR), is recommended for patients with CF. Aerobic exercise may help to mobilize secretions, in addition to providing the other known benefits of exercise in healthy individuals. Despite the benefits of PR programmes, low participant uptake, high drop-out rates, financial and transportation difficulties reduced the attendance in these programs. Different telemedicine treatments have been developed to overcome these difficulties and reduce healthcare costs. In recent studies, shows that tele-exercise is a promising new approach to promote exercise in children with CF. Although different exercise modalities such as aerobic exercise training and strength training have been investigated in CF patients, there is no study to examine stabilization exercises in this populations. Also there is no study to evaluate the effect of exercise training on irisin. In addition, although it is known that acute exercise has positive effects on both oxidant and antioxidant markers in the pediatric population, the effect of long-term exercise on oxidative stress has not been adequately studied. The aim of this study is to examine the effect of different exercise training modalities applied with telerehabilitation method on functional capacity, oxidative stress and respiratory parameters in CF patients. . In the study, after measuring respiratory functions, exercise capacity, oxidative stress parameters, peripheral muscle functions, balance, posture, quality of life and physical activity questionnaire, 39 people will be divided into three groups. First group will be applied only online supervised stabilization exercises, Second group will be applied online supervised aerobic exercise training and stabilization exercises. And the third group, the physical activity importance will be explained and appropriate physical activity recommendations will be made. All outcome measures will be repeated after exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 8-18 years with a diagnosis of cystic fibrosis (CF)
* Access to online exercise training
* Percent predicted of forced expiratory volume at one second (FEV1) > 40% in pulmonary function test

Exclusion Criteria:

* Being diagnosed with acute pulmonary exacerbation at the time of study and / or within the last month.
* Being physically or perceptually competent to exercise
* Patients with allergic bronchopulmonary aspergillosis (ABPA) who were treated with systemic steroid therapy
* Having FEV1 %< 40% at pulmonary function test.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
six minute walk test distance | before the exercise training
  Six-minute walk test distance is recorded
six minute walk test distance | eight week
  Six-minute walk test distance is recorded
shuttle walk test distance | before exercise training
  shuttle walk test distance is recorded
shuttle walk test distance | eight week
  shuttle walk test distance is recorded

SECONDARY OUTCOMES:
Respiratory muscle strength | before exercise training
  Respiratory muscle strength will be evaluated using mouth pressure device
Respiratory muscle strength | eight week
  Respiratory muscle strength will be evaluated using mouth pressure device
Respiratory muscle endurance | before exercise training
  Respiratory muscle endurance will be evaluated using constant load test
Respiratory muscle endurance | eight week
  Respiratory muscle endurance will be evaluated using constant load test
Pulmonary functions-FVC | before exercise training
  Forced vital capacity (FVC)
Pulmonary functions-FVC | eight week
  Forced vital capacity (FVC)
Pulmonary functions-FEV1 | before exercise training
  Forced expiratory volume in the first second (FEV1)
Pulmonary functions-FEV1 | eight week
  Forced expiratory volume in the first second (FEV1)
Pulmonary functions-FEV1/FVC | before exercise training
  FEV1/ FVC
Pulmonary functions-FEV1/FVC | eight week
  FEV1/ FVC
Pulmonary functions-PEF | before exercise training
  Peak Expiratory Flow (PEF)
Pulmonary functions-PEF | eight week
  Peak Expiratory Flow (PEF)
Pulmonary functions-FEF25-75 | before exercise training
  Forced mid-expiratory flow (FEF25-75)
Pulmonary functions-FEF25-75 | eight week
  Forced mid-expiratory flow (FEF25-75)
Oxidative stress-MDA | before exercise training
  Malondialdehyde (MDA) will be determined in the blood samples.
Oxidative stress-MDA | eight week
  Malondialdehyde (MDA) will be determined in the blood samples.
Oxidative stress-SOD | before exercise training
  Superoxide dismutase (SOD) will be determined in the blood samples.
Oxidative stress-SOD | eight week
  Superoxide dismutase (SOD) will be determined in the blood samples.
Oxidative stress-CAT | before exercise training
  Catalase (CAT) will be determined in the blood samples.
Oxidative stress-CAT | eight week
  Catalase (CAT) will be determined in the blood samples.
Oxidative stress-PC | before exercise training
  Protein carbonyl (PC) will be determined in the blood samples.
Oxidative stress-PC | eight week
  Protein carbonyl (PC) will be determined in the blood samples.
Oxidative stress-TOS | before exercise training
  Total oxidant status (TOS) will be determined in the blood samples.
Oxidative stress-TOS | eight week
  Total oxidant status (TOS) will be determined in the blood samples.
Oxidative stress-TAS | before exercise training
  Total antioxidant status(TAS) will be determined in the blood samples.
Oxidative stress-TAS | eight week
  Total antioxidant status (TAS) will be determined in the blood samples.
Oxidative stress-oxidative stress index | before exercise training
  Oxidative stress index (TOS/TAS)
Oxidative stress-oxidative stress index | eight week
  Oxidative stress index (TOS/TAS)
Peripheral muscle strength | before exercise training
  Peripheral muscle strength will be evaluated using dynamometer
Peripheral muscle strength | eight week
  Peripheral muscle strength will be evaluated using dynamometer
crunch repetitions | before exercise training
  number of crunch completed is recorded
crunch repetitions | eight week
  number of crunch completed is recorded
squat repetitions | before exercise training
  number of squats completed is recorded
squat repetitions | eight week
  number of squats completed is recorded
push-up repetitions | before exercise training
  number of push-ups completed is recorded
push-up repetitions | eight week
  number of push-ups completed is recorded
plank duration | before exercise training
  duration of keeping plank position is recorded
plank duration | eight week
  duration of keeping plank position is recorded
1 minute sit to stand test (STS) repetitions | before exercise training
  number of sit to stand for one minute is recorded
1 minute sit to stand test (STS) repetitions | eight week
  number of sit to stand for one minute is recorded
myokine assessment | before exercise training
  irisin levels will be determined in the blood sample
myokine assessment | eight week
  irisin levels will be determined in the blood sample
posture-Corbin | before exercise training
  Posture will be evaluated using Corbin Postural Assessment scale. Lateral and posterior views will be assessed (0 = absent, 1 = mild, 2 = moderate, 3 = severe) and posture score will be determined as excellent (0-2), very good (3-4), good (5-7), fair (8-11) and poor (>12).
posture-Corbin | eight week
  Posture will be evaluated using Corbin Postural Assessment scale. Lateral and posterior views will be assessed (0 = absent, 1 = mild, 2 = moderate, 3 = severe) and posture score will be determined as excellent (0-2), very good (3-4), good (5-7), fair (8-11) and poor (>12).
posture | before exercise training
  Thoracic kyphosis and lumbar lordosis angles will be evaluated in the sagittal plane with spinal mouse device.
posture | eight week
  Thoracic kyphosis and lumbar lordosis angles will be evaluated in the sagittal plane with spinal mouse device.
balance | before exercise training
  Pediatric berg balance scale will be used. The scale consists of 14 parts. Each section is scored between 0-4. The highest score that can be obtained from the scale is 56.Higher score means a better outcome.
balance | eight week
  Pediatric berg balance scale will be used. The scale consists of 14 parts. Each section is scored between 0-4. The highest score that can be obtained from the scale is 56.Higher score means a better outcome.
static balance | before exercise training
  static balance will be evaluated functional reach test
static balance | eight week
  static balance will be evaluated functional reach test
dynamic balance | before exercise training
  Balance will be evaluated using one-legged standing test
dynamic balance | eight week
  Balance will be evaluated using one-legged standing test
functional mobility | before exercise training
  functional mobility will be evaluated time-up go test
functional mobility | eight week
  functional mobility will be evaluated time-up go test
Mcgill core endurance test | before exercise training
  Endurance of trunk muscles will be evaluated trunk flexor, trunk extensor and side plank test
Mcgill core endurance test | eight week
  Endurance of trunk muscles will be evaluated trunk flexor, trunk extensor and side plank test
Quality of life assessment | before exercise training
  Quality of life will be evaluated using the Cystic Fibrosis Questionnaire-Revised (CFQ-R).The Cystic Fibrosis Questionnaire-Revised (CFQ-R) is a disease-specific health-related quality of life (HRQOL) measure for children, adolescents with cystic fibrosis (CF). The questionnaire assess physical functioning, emotional functioning, social functioning, body image, eating disorders, treatment, respiratory symptoms and digestive symptoms.Score range is 0-100. Higher scores indicating higher health-related quality of life.
Quality of life assessment | eight week
  Quality of life will be evaluated using the Cystic Fibrosis Questionnaire-Revised (CFQ-R).The Cystic Fibrosis Questionnaire-Revised (CFQ-R) is a disease-specific health-related quality of life (HRQOL) measure for children, adolescents with cystic fibrosis (CF). The questionnaire assess physical functioning, emotional functioning, social functioning, body image, eating disorders, treatment, respiratory symptoms and digestive symptoms.Score range is 0-100. Higher scores indicating higher health-related quality of life.
Physical activity assessment | before exercise training
  Physical activity levels will be assessed by The Physical Activity Questionnaire. Score range is 1-5. Higher scores indicating higher physical activity
Physical activity assessment | eight week
  Physical activity levels will be assessed by The Physical Activity Questionnaire. Score range is 1-5. Higher scores indicating higher physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Dogru-Ersoz, Professor, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)